CLINICAL TRIAL: NCT02695784
Title: Probiotics After Discharge (PAD) Study: Impact on Microbiome, Health and Growth Outcomes
Brief Title: Probiotics After Discharge
Acronym: PAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7840
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Microbiota; Bacteriophages; Infantile Colic; Growth
MeSH Terms: conditions — Colic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic continuation (Experimental): This Group will Continue probiotics Beyond 34 weeks corrected Gestational agent standard practice
  Interventions: Dietary Supplement: Probiotic Continuation
- Standard treatment Group (No Intervention): This group will continue current standard practice of stopping probiotics at 34 weeks corrected gestational age

INTERVENTIONS:
Dietary Supplement: Probiotic Continuation — This arm will continue to receive probiotics beyond 34 weeks corrected gestation until two months after discharge
  Arms: Probiotic continuation

SUMMARY:
The influence of the preterm gut microbiota in health and disease has been well established. However, relatively little is known about how the microbiome changes after discharge and its relationship with growth, health and disease outcomes in the preterm population. This study aims to follow a cohort of preterm infants and explore the relationship of the later microbiome ('after discharge') with later growth and health outcomes in infancy. The study will also explore the effect of timing of stopping routinely administered probiotics on the post-discharge microbiome, infant feeding and outcomes such as colic.

The investigators aim to longitudinally follow 40 infants born before 32 weeks gestation who have also taken part in the investigators microbiome study during their NICU stay (SERVIS REC No: 10/H0908/39) and where microbiomic sampling has been adequately achieved. The investigators will collect stool at and beyond the time of anticipated discharge (beyond 34 weeks) targeted to include pre- and post-weaning, and again at a year. Actual discharge timing of these infants varies, and is usually latest in the most immature infants, allowing an assessment of the influence of physical location (NICU vs home) as well as increasing age. Using 16S ribosomal RNA amplicon analysis, the investigators will assess bacterial colonisation of the gut and measure infant weight, length and head circumference at each time point. The investigators will use a parent questionnaire to assess daily crying time, parents' perceptions of colic severity using a visual analogue scale as well as vomiting and constipation for the two weeks before sampling.

ELIGIBILITY:
Inclusion Criteria:

* <32 weeks Corrected Gestation
* Followed up in Newcastle Region

Exclusion Criteria:

-

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome | one year
  16S RNA assessed using illumina sequencer

SECONDARY OUTCOMES:
Growth Velocity | 1 year
  Weight Increase in g/kg/day
Head Growth | 1 year
  cm/kg/day
Growth: Length | 1 year
  Length: cm/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Janet Berrington, Principal Investigator — Newcastle NHS FOundation Trust
Locations (1):
- Newcastle Neonatal Service, Newcastle upon Tyne, Tyne and Wear, United Kingdom